CLINICAL TRIAL: NCT04063657
Title: External Fixation Versus Splinting of Acute Calcaneus Fractures Prior to Definitive Surgery
Brief Title: External Fixation Versus Splinting of Acute Calcaneus Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was slow to recruit. PI decided to close study to focus on other trials.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1436830
Record Dates: First submitted 2019-08-07; First posted 2019-08-21 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Calcaneus Fracture
Keywords: Staged External Fixation; Splinting; Soft tissue complications
MeSH Terms: interventions — External Fixators; Splints

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- External fixation (Active Comparator): Adults diagnosed with an acute (<2 days from injury) calcaneal fracture recommended for operative treatment will be placed in external fixator until the patient is deemed clinically appropriate for definitive surgical fixation.
  Interventions: Procedure: External fixator
- Splinting (Active Comparator): Adults diagnosed with an acute (<2 days from injury) calcaneal fracture recommended for operative treatment will be placed in a short leg splint until the patient is deemed clinically appropriate for definitive surgical fixation.
  Interventions: Procedure: Splinting

INTERVENTIONS:
Procedure: External fixator — Patients will be placed in an external fixator followed by open versus closed surgical stabilization of their calcaneus fracture when their soft tissue is appropriate for surgery.
  Arms: External fixation
Procedure: Splinting — Patients will be placed in a short leg splint followed by open versus closed surgical stabilization of their calcaneus fracture when their soft tissue is appropriate for surgery.
  Arms: Splinting

SUMMARY:
Aim:

* Determine if external fixation decreases soft tissue complications compared to splinting.
* Determine if external fixation decreases time to definitive surgical stabilization and improves final fixation compared to splinting.
* Determine if external fixation improves functional outcomes as evaluated by validated functional scoring systems.

Hypothesis:

* External fixation improves definitive fixation and functional outcomes of acute calcaneal fractures with decreased complication rates compared to splinting

ELIGIBILITY:
Inclusion Criteria:

* Voluntary consent
* Age 18 to 69
* Clinical and/or advanced imaging confirming an acute calcaneal fracture that has occurred within 2 days of which, eventually definitive surgery is recommended/accepted.
* Unable to consent

Exclusion Criteria:

* Age <18
* Prior surgery of the affected extremity
* Prisoners
* Pregnant women
* Inflammatory arthritis
* Non-English-speaking patients

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Kreulen, MD, MS, Principal Investigator — Foot and Ankle Surgery Department of Orthopaedic Surgery University of California, Davis Medical Center
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | External Fixation | Splinting
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study stopped prematurely, only 1 participant enrolled in the external fixation arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | External Fixation | Splinting | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 50 [50 to 50] |  | 50 [50 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 0 |  | 0
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Definitive Surgery
Description: Duration of time from injury to definitive surgery
Time Frame: Within 2 weeks from injury
Population: Study stopped prematurely due to poor recruitment. Only 1 subject was enrolled.
Measure: Number; unit: days
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 1 | 0
days | 3 |

2. Primary Outcome: Soft Tissue Complications
Description: Incidence of infection, dehiscence and need for soft tissue coverage
Time Frame: Assessed at 2 weeks after surgery
Population: Study stopped prematurely due to poor recruitment. Only 1 participant was enrolled. Participant did not attend follow up visit where this data would have been collected.
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Soft Tissue Complications
Description: Incidence of infection, dehiscence and need for soft tissue coverage
Time Frame: Assessed at 6 weeks after surgery
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Soft Tissue Complications
Description: Incidence of infection, dehiscence and need for soft tissue coverage
Time Frame: Assessed at 12 weeks after surgery
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Soft Tissue Complications
Description: Incidence of infection, dehiscence and need for soft tissue coverage
Time Frame: Assessed at 6 months after surgery
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Soft Tissue Complications
Description: Incidence of infection, dehiscence and need for soft tissue coverage
Time Frame: Assessed at 12 months after surgery
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Soft Tissue Complications
Description: Incidence of infection, dehiscence and need for soft tissue coverage
Time Frame: Assessed at 24 months after surgery
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Union Rate
Description: Assessment of fracture healing
Time Frame: Plain xrays at 6 weeks, 12 weeks, 6 months, 1 year, and 2 years after surgery. CT scan at 1 year.
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Radiographic Parameters - Bohler's Angle
Description: Bohler's angle
Time Frame: Assessed at 2, 6, & 12 weeks, and 6, 12, & 24 months after surgery
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Radiographic Parameters - Calcaneal Height
Description: Calcaneal height
Time Frame: Assessed at 2, 6, & 12 weeks, and 6, 12, & 24 months after surgery
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Radiographic Parameters - Angle of Gissan
Description: Angle of Gissan
Time Frame: Assessed at 2, 6, & 12 weeks, and 6, 12, & 24 months after surgery
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Radiographic Parameters - Calcaneal Width
Description: Calcaneal width
Time Frame: Assessed at 2, 6, & 12 weeks, and 6, 12, & 24 months after surgery
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Radiographic Parameters - Calcaneal Length
Description: Calcaneal length
Time Frame: Assessed at 2, 6, & 12 weeks, and 6, 12, & 24 months after surgery
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Functional Outcomes - VAS
Description: Assess Visual Analogue pain score(VAS). This will be a patient reported measure from 0-10, minimum score of 0 (no pain), maximum score of 10 (most pain).
Time Frame: Assessed at 2, 6, & 12 weeks, and 6, 12, & 24 months after surgery.
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Functional Outcomes - FFI-R
Description: Revised foot function index questionnaire (FFI-R) will assess patient pain, stiffness, activity, difficulties with ambulation, and social issues. The score is tabulated from 34 questions answered 1-5 (1= none of the time, 5= All of the time, scale 34-170). Higher scores indicate worse outcomes.
Time Frame: Assessed at 2, 6, & 12 weeks, and 6, 12, & 24 months after surgery
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Functional Outcomes - FAAM ADL
Description: Foot and Ankle Ability measure activities of daily living (FAAM ADL) is a 21-item activities assessing the patient's functionality related to their activities of daily living. The response to each item is scored from 4 to 0, with 4 being ''no difficulty'' and 0 being ''unable to do." Scale 0-84. Higher scores indicate a more favorable functional level.
Time Frame: Assessed at 2, 6, & 12 weeks, and 6, 12, & 24 months after surgery
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Functional Outcomes - FAAM Sport
Description: Foot and Ankle Ability measure activities of daily living (FAAM Sport) is a 8-item questionnaire assess the patient's ability to participate in athletic activities. The response to each item is scored from 4 to 0, with 4 being ''no difficulty'' and 0 being ''unable to do." Scale 0-32. Higher scores indicate a more favorable functional level.
Time Frame: Assessed at 2, 6, & 12 weeks, and 6, 12, & 24 months after surgery
Population: as for outcome 2
Arm/Group | External Fixation | Splinting
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: Study stopped prematurely due to poor recruitment. Only 1 participant was enrolled. Participant was lost to follow-up and did not attend follow up visits.
Arm/Group | External Fixation | Splinting
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Study stopped prematurely due to poor recruitment. Only 1 participant was enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT04063657/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT04063657/ICF_001.pdf